

# Subject information for participation for medical-scientific research

# Comparing two different surgical techniques to remove the womb via the vagina

Vaginal hysterectomy versus vaginally-Assisted NOTES Hysterectomy (VANH): a randomised controlled trial (VANH-trial)

### Introduction

Dear madam,

In this information letter you will find information about medical-scientific research. Participating in this research is voluntary. You receive this letter because you will get an operation to remove the uterus vaginally.

In this letter you will receive information about what kind of research this is, what is means for you, and what the advantages and disadvantages are. Would you please read this information and decide whether you want to participate? If you want to participate, kindly fill out the form in attachment E.

### Ask your questions

You can take your decision with the information that you can find in this information letter. Next to this, we advise you to do the following:

- Ask questions to the investigator who gives you this information.
- Talk to your partner, family or friends about this research.
- Ask questions to the independent expert, Dr. R. Hendrickx.
- Read information at www.rijksoverheid.nl/mensenonderzoek.

# 1. General information

Zuyderland Medical Centre, department of Gynecology, started this research. From now on, Zuyderland Medical Centre will be called 'client'. Investigators (doctors) perform this study in different hospitals. For this research, a total of 124 patients is necessary from different hospitals. The Medical-Ethic research Committee Zuyderland (METC Z) approved this research.

VANH-trial, patient informationfolder, version 2, 13-03-2021

2. What is the goal of this research?

Since hundreds of years, the uterus has been removed through the vagina. Other ways to remove the

uterus are with using a laparoscopy or with a cut in the under-abdomen.

Since a couple of years, a new technique has been introduced, the vNOTES technique, wherein the

uterus is removed vaginally using endoscopy. The abbreviation vNOTES stands for vaginal Natural

Orifice Transluminal Endoscopic surgery, which means that natural orifices (for example the vagina)

are used to perform endoscopic surgery.

Former research has shown that removing the uterus with the vNOTES technique seems as good as

removing the uterus endoscopically.

The goal of the research is to compare two ways to remove the uterus vaginally, via the original

vaginal route or by using the vNOTES technique.

3. What is the background of the research?

The removal of the uterus is possible in different ways. Every technique has its pros and cons. We

want to investigate whether the removal of the uterus by the vNOTES technique gives less pain

compared to the normal vaginal route. Less pain means less use of pain medication after surgery and

even a quicker discharge after surgery.

4. How elapses the research?

How long does the research take?

Are you participating in the study? Than this will take about 6 weeks. This is as long as the normal

recovery period after vaginally removing of the uterus.

Step 1: are you suited to participate?

First, we want to be sure that you are suitable to participate. The investigator will do a research:

• Physical gynecological examination

• Research to your medical history and medication use

Step 2: the treatment/ the surgery

For this research we will make 2 groups:

Group 1. The people in this group will get the surgery using the vNOTES technique

2

• Group 2. The people in this group will get the surgery using the conventional vaginal technique.

It will be randomly be decided which group you will get in to. You don't know in which surgery you will undergo. If this is necessary to know for your general health, this can be made public. When the research has finished, we will let you know which surgery you have had.

### Step 3: research and measurements

For this research, it is not necessary to make extra visits to the hospital. Six to eight weeks after surgery, you will have a hospital visit for standard control. We do ask you to fill in (extra) questionnaires.

We will do the following examinations:

- Physical gynaecological examination.
- You will fill in questionnaires. The questions are about general information, complaints of pain before and after the surgery and recovery after surgery.

Attachments C consists of the measurements that we will perform with every visit and how often you will receive a questionnaire.

We will send you a questionnaire about 3-4 times.

The questions will go about the recovery after the surgery. It will take about 5-10 minutes each time to fill in the questionnaire.

# Step 4: follow-up

In this study, the follow-up is not different compared to the normal care. The follow-up appointments are the same as the appointments that you would have had after surgery without the study.

### 5. Which agreements will we make?

We want the study to go fluently. That is why we will make the next agreements with you:

- You will not participate in other medical research without first consulting the investigators of this study first.
- You will come to each appointment.
- You will fill in the questionnaire before and after the surgery.

You will get in touch with the investigators in the next situations:

- You are being admitted or treated in the hospital
- You suddenly experience health issues
- You don't want to participate in the study anymore
- Your phone number, address or email-address has been changed.

Can you get pregnant during this study?

Women who are pregnant, cannot participate in this study.

Getting pregnant after the study?

It is not possible anymore to get pregnant after you have participated in this study, because your uterus has been removed.

# 6. What side-effects, negative effects or inconveniences can you get of participating?

The vNOTES surgical technique probably has no additional risks or side-effects compared to the conventional vaginal hysterectomy.

## 7. What are the pros and cons of participating in the study?

Participating in the study can have pros and cos. These are high lighted below. Think about this very carefully and talk about the study with others.

Participating in the study can have the following pros:

We think that the vaginal hysterectomy using the vNOTES technique gives less pain after the surgery, but this is not a certainty. Because the investigators think that less pain is experienced, they also think that it is more often possible to be discharged from the hospital at the day of the surgery.

Participating in the study can have the following cons:

You are not freely to choose which surgery you will receive, but this will be randomly chosen.

The questionnaires will take about 30-60 minutes of you time.

You do not want to participate?

Participating in the study is voluntary, you decide yourself whether you want to participate or not. When you do not want to participate in the study, you will get the conventional treatment to remove your uterus. Your doctor can tell you more about the different methods end the pros and cons of each method.

# 8. When does the study stop?

The investigator will keep you posted when they have new information which is important for you. The investigator will ask you again after given this information if you still want to participate. In the following situations the study will stop for you:

- All examinations according to the schedule are over.
- You want to stop participating in the study. You can leave the study at any moment. Tell this
  to the investigator when you want to stop. You are not obligated to give a reason. You will
  receive the regular treatment for removing the uterus. The investigator will invite you for the
  follow-up.
- The investigator thinks it is better for you to stop participating. He or she will invite you for the follow-up appointment.
- One of the following organizations thinks it is better to stop the study:
  - o The department of Gynecology and Obstetrics Zuyderland Medical Centre
  - The government
  - The Medical Ethical committee (METC-Z) who is assessing the study.

What will happen when you stop participating?

The investigators will use the data that already has been collected before stopping participation. The study is finished when all participants completed the examinations.

## 9. What will happen after the study?

Will you get the results of the study?

In about 1-2 years after your participation, the investigators will let you know what the most important results of the study are. The investigator can also let you know which surgery you have had. When you don't want to know this information, you can tell your investigator. They will then not inform you.

### 10. What will we be doing with your data?

Are participating in the study? Then you also give permission to collect, use and save your data

Which data do we save?

We save the following data:

- Your name
- Your sex
- Your address
- Your birthdate
- Information about your health
- (Medical) information that we collect during the study

Why do we collect, use and save your data?

We collect, use and save your data to be able to answer the question in this study and to publish the results.

How do we protect your privacy?

To protect your privacy, we will give your data a code. All your data will receive this code. The key of this code will be saved on a save spot in the hospital. When we use your data, only the code will be used. In publications or reports it is not possible to recall which data is yours.

Who is able to see your data?

Some people are allowed to know your name and other personal information without the code. These are the people who control the investigators whether they are preforming the study in a save and reliable way. The people who can see these data are:

- Committee who is keeping an eye on the safety of the study.
- A supervisor who has been hired by the Zuyderland Medical Centre.
- National and international authorities, for example the inspection of public health and youth.

These people will keep your data private. We will ask your permission for insight in this information.

How long do we save your data?

We will save your data for 15 years in the hospital and 15 years with the client.

#### Can we have your data?

Your data can also be important for research after completing this study, to improve the new method. This is why your data will be saved for 15 years in the hospital. In this form, you can give your permission. Do you not want to give your permission? Than it is still possible to participate in the study, and you will receive the same care.

What happens when something unexpected occurs?

It is possible that we will find something during the study that is important for your health. The investigator will then get in contact with your general practicer. You will talk to your GP or specialist what to do next. You can give your permission for informing your GP.

Is is possible to take back your permission for using your data?

It is possible to take back your permission at any moment. This applies for the permission for this study only as well as the permission to use your data in other research. But be aware, do you stop giving permission and did the investigators already retrieve some? Then they are allowed to use that data.

Do you want to know more about your privacy?

- Do you want to know more about your rights with using your personal data? You can check the following website: <a href="https://www.autoriteitpersoonsgegevens.nl">www.autoriteitpersoonsgegevens.nl</a>.
- Do you have questions about your rights? Or do you have a complaint about using your personal data? Get in contact with the person who is responsible for the use of your personal data. For this study this is: see attachment A for contact information and the website.
- If you have complaints about the processing of your data, we advise you to first consult the investigation team. You can also consult the 'Functionaris Gegevensbescherming' of the Zuyderland Medical Centre. You can also file a complaint at the 'Autoriteit Persoonsgegevens'.

Where can you find more information about the study?

On the following website you can find more information about the study; <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a>. After the study, this website can give you a summary and the results of the study. You can find the study by searching for 'VANH-trial'.

#### 11. Do you get compensation for participating in the study?

The treatment for the study is for free, the surgery will be paid by your insurance. You do not get any compensation for participating in the study.

# 12. Are you insured during the study?

Everyone who is participating is insured through the study. The insurance will pay for any damage due to the study, but not for all damage. In **attachment B**, you will find more information about the insurance and exceptions. Here you will also find information about where to claim your damage.

### 13. We inform your GP

The investigator will send a letter to your GP to let them know that you are participating in the study. This is for your own safety.

#### 14. Do you have any questions?

Questions about the study can you ask at the research team. Do you want any advice from someone who doesn't have any interest in the study? Then you can go to dr. R. Hendrickx. He knows a lot about the study, but is not participating in the study.

Do you have a complaint? You can discuss this with the investigator or your doctor. Would you rather not consult them? Then you can get in touch with the complaints officer of the Zuyderland Medical Centre. Attachment A contains contact information.

### 15. How do you give consent for participation in this study?

You can take your time to carefully think about participating in this study. Your lawful reflection period is 7 days. After these 7 days you can tell the researcher whether you understand the information and if you want to participate or not. Would you like to participate? Then you can fill in the consent form that you will find together with this information letter. You and the researcher will both receive a signed version of this consent form. Would you not like to participate? If you rather not like to participate in this study, we would like to ask you if it is a problem to collect your data without you having to complete an operation or questionnaires. The separate consent form to collect your data for this study is called "cohort".

Thanks for your time.

#### 16. Attachment of this information folder

- A. Contact details Zuyderland Medical Center
- B. Insurance information
- C. Schedule of research measurements
- D. Information about possible side effects
- E. VANH trial consent forms
- F. Consent forms Cohort

### **Attachment A: Contact details Zuyderland Medical Centre**

#### Research team:

Name: Dr. M.M.L.H. Wassen

Function: Gynecologist, Obstetrics and Gynecology

Contact details: m.wassen@zuyderland.nl

Availability: Monday-Sunday from 08:00am to 5:00pm.

Name: I.P.W. Bekkers

Function: Resident Gynecology and Obstetrics

Contact details: il.bekkers@zuyderland.nl

Availability: Monday-Sunday from 8:00am to 5:00pm.

Independent physician: dr. R. Hendrickx

Function: Orthopedic surgeon Zuyderland Medical Centre

Contact details: r.hendrickx@zuyderland.nl

#### **Complaints**

If you have any complaints about this research you can report this to the researchers. When you prefer not do this you can contact the Patient Service Bureau Zuyderland, phone number: 088-4596300.

# More information about you rights when processing your data

For general information about your rights when processing your personal data you can consult the website of the Dutch Data Protection Authority. If you have any questions or complaints about the

VANH-trial, patient informationfolder, version 2, 13-03-2021

use or processing of your data or about your rights please contact the Data Protection Officer (DPO)

of Zuyderland Medical Center: Name: Mrs. Marianne Korpershoek; Telephone number: 088-45 97

777; Email: <a href="mailto:privacy@zuderland.nl">privacy@zuderland.nl</a>; link to privacy statements/privacy regulations of Zuyderland:

https://www.zuyderland.nl/wp-content/uploads/2016/06/Privacyreglement-t.b.v.-Zuyderland:

patiëntgegevens.pdf

Attachment B: Information about the insurance

Zuyderland Medical Center has an insurance for everyone participating in the study. The insurance

pays for the damage you have sustained by participating in this study. This concerns damage you

have sustained during the study or within 4 years after the study. You must report this damage to the

insurance company within 4 years.

Did you suffer damage as a result of this study? Report this to the insurance company:

You can contact the insurance company by telephone as described below.

The insurance company of the study is:

Name: Onderlinge Waarborgmaatschappij Centramed

Address: Maria Montessorilaan 9, 2719DB, Zoetermeer

Telephone number: 070-3017070

E-mail: info@centramed.nl

Policy number: 624.455.607

De verzekering betaalt maximaal € 650.000 per persoon en € 5.000.000 voor het hele onderzoek €

7.500.000 per jaar voor alle onderzoeken van dezelfde opdrachtgever.

The insurance pays a maximum of €650.000 per person and €5.000.000 for the entire study and

€7.500.000 per year for all the studies of the same assigning party.

Please note: the insurance **does not** cover the following damage:

• Damage due to a risk about which we have informed you in this letter. But this does not

apply when the risk turned out to be greater than we previously thought. Or if the risk was

very unlikely.

Damage to your health that would also have occurred if you would have not participated in

this study.

Damage that arises because you did not follow directions or instructions properly.

10

- Damage to the health of your children or grandchildren.
- Damage due to a treatment method that already exists. Or through research into a treatment method that already exists.

These provisions are stated in the 'Besluit verplichte verzekering bij medisch-wetenschappelijk onderzoek met mensen 2015'. This statement can be found in the government's overview of laws (https://wetten.overheid.nl).

#### **Attachment C: Schedule of research measurements**

Below is the diagram in which the measurements are displayed. The different moments of measurements are listed in the left column. The columns on the right (consent (basic), questionnaire and pain score) show when you will receive the different questions. This is marked by a blue box.

| | Consent | Basic<br>questionnaire | Questionnaire after the surgery | Pain score |
|---|---|---|---|---|
| Outpatient clinic visit | | | | |
| Start of the investigation | | | | |
| 1 hour after the surgery | | | | |
| 8 hours after the surgery | | | | |
| 24 hours after the surgery (at home or at the ward) | | | | |
| Day 2-7 after the surgery (Online and on | | | | |

| paper) |
|-----------------------------------------------------|
| 4 weeks after the surgery (online) |
| 6 weeks after the surgery (outpatient clinic visit) |
| 12 weeks after the surgery (online) |

# Attachment D – Side effect, adverse effects and discomforts

The study does not indicate a higher risk of complications or side effects compared to normal vaginal removal of the uterus.

# Attachment E: consent form trial subject

Belonging to the VANH-trial:

- I have read the information letter. I had the possibility to ask questions. My questions have been answered well enough. I had enough time to decide whether I would like to participate.
- I am aware that participation is voluntary. I know that I can decide at any time to not participate in the study anymore or to quit. I know that I do not need to mention the reason why I want to quit.
- I give the researcher my permission to inform my GP that I am participating in this study.
- I give the researcher permission to provide my GP or specialist with information about unexpected findings from the research that is important for my health.
- I give the researchers permission to collect and use my data. The researchers only use this data for the sake of interest to answer the research question of this study.
- I am aware that some people will be able to view all of my data for the verification of the study. Those people are mentioned in this information letter. I give these people permission to view my data for this verification.
- I know that I cannot be pregnant during the study.
- The researcher discussed with me how I can prevent getting pregnant.

Do you want to choose yes or no in the table below?

| I give permission to save my data in order to use it for other | Yes □ | No □ |
|---|---|---|
| research, as stated in the information letter. | | |
| I give permission to ask me if I want to participate in a | Yes □ | No □ |
| follow-up study after this study. | | |
| I give the researchers permission to let me know which | Yes 🗆 | No □ |
| treatment I received/in which group I was after the study. | | |

Signature:....

The trial subject will receive a complete information letter together with a signed version of the consent form.

Date: \_\_ / \_\_ / \_\_

# Attachment F: consent form trial subject

Belonging to the cohort:

- I have read the information letter. I had the possibility to ask questions. My questions have been answered well enough. I had enough time to decide whether I would like to participate.
- I am aware that participation is voluntary. I know that I can decide at any time to not participate in the study anymore or to quit. I know that I do not need to mention the reason why I want to quit.
- I give the researcher my permission to inform my GP that I am participating in this study.
- I give the researcher permission to provide my GP or specialist with information about unexpected findings from the research that is important for my health.
- I give the researchers permission to collect and use my data. The researchers only use this data for the sake of interest to answer the research question of this study.
- I am aware that some people will be able to view all of my data for the verification of the study. Those people are mentioned in this information letter. I give these people permission to view my data for this verification.
- I know that I cannot be pregnant during the study.
- The researcher discussed with me how I can prevent getting pregnant.

Do you want to choose yes or no in the table below?

| I give permission to save my data in order to use it for other | Yes □ | No□ |
|----------------------------------------------------------------|-------|-----|
| research, as stated in the information letter. | | |
| I give permission to ask me if I want to participate in a | Yes □ | No□ |
| follow-up study after this study. | | |
| I give the researchers permission to let me know which | Yes 🗆 | No□ |
| treatment I received/in which group I was after the study. | | |

• I want to participate in this study.

| My name is (trial subject): | | |
|-----------------------------|------|--------|
| Signature: | Date | :_/_/_ |

VANH-trial, patient informationfolder, version 2, 13-03-2021

I declare that I have fully informed the trial subject about the mentioned study.

If during the study any information will be known that could influence the subject's consent? Then I will let the trial subject know this in time.

| Name researcher (or its representative): | |
|------------------------------------------|-----------|
| Signature: | Date: / / |
| Additional information is provided by: | |
| Name: | |
| Function: | |
| Signature: | Date: / / |

The trial subject will receive a complete information letter together with a signed version of the consent form.